CLINICAL TRIAL: NCT02378077
Title: Immunomodulatory Role of Eosinophils in Determining Inflammation and Insulin Sensitivity in Human Adipose Tissue- Aims 1&2
Brief Title: Understanding the Relationship Between Inflammation and Insulin Resistance in the Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elena Anna (Eleanna) De Filippis, M.D., Ph.D., Senior Consultant of Endocrinology and Metabolic Disease, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-001288
Record Dates: First submitted 2014-09-17; First posted 2015-03-04 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean or Obese, Non-Diabetic (Experimental): To determine whether eosinophil content of adipose tissue is related to insulin sensitivity. We will use euglycemic clamps, fat biopsy (obtained during a scheduled abdominal surgery) and fat aspiration for analysis of subcutaneous (Sc) and omental (OM) adipose tissue from obese, insulin resistant and lean, insulin sensitive volunteers to test the hypothesis that, as in mice, eosinophil content in human subcutaneous and omental white adipose tissue, inversely correlates with body weight, with skeletal muscle and hepatic insulin sensitivity.
  Interventions: Procedure: Fat biopsy during scheduled abdominal surgery; Procedure: Fat Aspiration
- Fish oil supplementation (Experimental): Determine whether, in adipose tissue, levels of, anti-inflammatory molecules correlate with insulin sensitivity and whether these levels are altered by a treatment designed to promote resolution of inflammation. Volunteers will take a fish oil supplement for three months.
  Interventions: Procedure: Fat Aspiration; Dietary Supplement: Fish Oil Supplement

INTERVENTIONS:
Procedure: Fat biopsy during scheduled abdominal surgery — Physical exam including blood work, an EKG and bioimpedance testing. An oral glucose tolerance test. Insulin infusion. Fat tissue biopsy during a scheduled abdominal surgery.
  Other Names: Fat Aspiration; Tissue Biopsy
  Arms: Lean or Obese, Non-Diabetic
Procedure: Fat Aspiration — Physical exam including blood work, an EKG and bioimpedance testing. An oral glucose tolerance test. Insulin infusion. Subcutaneous fat tissue biopsy.
  Other Names: Fat Sample; Adipose Tissue
Dietary Supplement: Fish Oil Supplement — Fish Oil supplementation for three months.
  Other Names: Dietary Supplement
  Arms: Fish oil supplementation

SUMMARY:
This study is being done to better understand the relationship between inflammation and insulin resistance in your Adipose (fat) Tissue .

DETAILED DESCRIPTION:
This study is being done to determine whether eosinophils (a type of white blood cell) play an important role in human fat metabolism and inflammation.

This study is being done to determine if fish oil supplement could play a role in reducing inflammation and improving insulin sensitivity in your fat tissue.

ELIGIBILITY:
Lean, healthy person with a body mass index (BMI) of 25 or less, or you are obese, BMI between 30 and 50, and non-diabetic.

Lean healthy controls will not be on any medication and will be undergoing elective abdominal surgery excluding those involving acute inflammation (i.e. acute cholecystitis, bowel perforation, or diverticulitis).

Obese, non-diabetic subjects will have a BMI between 30 and 50 and be taking no medications affecting glucose metabolism or lipid metabolism. These subjects will be identified from a pool of patients undergoing an elective abdominal surgical procedure such as inguinal hernia repair, laparoscopic Nissen fundoplication, planned cholecystectomy, but also bariatric surgery.

Volunteers will not be taking corticosteroid therapy or have a history of asthma, COPD or atopic syndrome. All subjects will undergo a medical history intake and a physical examination followed by an OGTT to confirm normal glucose.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Eosinophil content in adipose tissue | baseline
  Eosinophils number will be measured by flow cytometry in subcutaneous and visceral fat of lean vs obese, non-diabetic volunteers

SECONDARY OUTCOMES:
Relationship between eosinophils content and body mass index (BMI) | baseline
  Measure as a linear regression between BMI (kg/m2) and eosinophils number in the fat

OTHER OUTCOMES:
Change in insulin sensitivity | Baseline, post fish oil supplementation (approximately 3 months)
  Measured by euglycemic-hyperinsulinemic clamp taken before and after fish oil supplementation
Change in plasma inflammatory cytokines | Baseline, post fish oil supplementation (approximately 3 months)
  Measured by Elisa reported in pg/mL before and after fish oil supplementation
Change in plasma inflammatory adipokines | Baseline, post fish oil supplementation (approximately 3 months)
  Measured by Elisa reported in pg/mL before and after fish oil supplementation
Change in adipose tissue inflammatory markers | Baseline, post fish oil supplementation (approximately 3 months)
  Measured by mRNA levels of pro-inflammatory markers before and after fish oil supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Elena Anna De Filippis, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Hernandez JD, Li T, Ghannam H, Rau CM, Masuda MY, Madura JA 2nd, Jacobsen EA, De Filippis E. Linking adipose tissue eosinophils, IL-4, and leptin in human obesity and insulin resistance. JCI Insight. 2024 Feb 8;9(3):e170772. doi: 10.1172/jci.insight.170772. PMID 38206766
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials